CLINICAL TRIAL: NCT03440697
Title: Pathogenetic Basis of Aortopathy and Aortic Valve Disease
Acronym: TAA
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Benjamin Landis, Associate Professor of Pediatrics, Indiana University
Other Study IDs: 1509977311
Record Dates: First submitted 2017-10-06; First posted 2018-02-22 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Aortopathies; Thoracic Aortic Aneurysm; Aortic Valve Disease; Thoracic Aortic Disease; Thoracic Aortic Dissection; Thoracic Aortic Rupture; Ascending Aortic Disease; Descending Aortic Disease; Ascending Aortic Aneurysm; Descending Aortic Aneurysm; Marfan Syndrome; Loeys-Dietz Syndrome; Vascular Ehlers-Danlos Syndrome; Shprintzen-Goldberg Syndrome; Turner Syndrome; PHACE Syndrome; Autosomal Recessive Cutis Laxa; Congenital Contractural Arachnodactyly; Arterial Tortuosity Syndrome; Bicuspid Aortic Valve-Associated Aortopathy; Bicuspid Aortic Valve; Familial Thoracic Aortic Aneurysm and Aortic Dissection
Keywords: Cardiac Disease; Cardiovascular Genetics
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Valve Disease; Dissection, Thoracic Aorta; Aneurysm, Ascending Aorta; Marfan Syndrome; Loeys-Dietz Syndrome; Ehlers-Danlos Syndrome, Type IV; Shprintzen Golberg craniosynostosis; Turner Syndrome; Aortic Aneurysm, Giant Congenital; Cutis Laxa, Autosomal Recessive, Type I; Congenital contractural arachnodactyly; Arterial Tortuosity Syndrome; Bicuspid Aortic Valve Disease; Aortic Aneurysm, Familial Thoracic 1; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Tissue, Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Aortopathy- Closed to external enrollment: Subjects with aortic disease including TAA or dissection, aortic tortuosity, or aortic hypoplasia/stenosis (based on any cardiac imaging modality including echocardiography, CT, MRI, or angiography)
- Syndromic- Open to external enrollment: Subjects with a genetic diagnosis of Marfan Syndrome (MFS), Loeys-Dietz Syndrome (LDS), Vascular Ehlers-Danlos Syndrome (EDS)
  •positive genetic testing and/or a previous cardiac study required to be eligible
- Aortopathy with Positive Genetic Results- Open to Enrollment: Subjects with aortic disease including TAA or dissection, aortic tortuosity, or aortic hypoplasia/stenosis (based on any cardiac imaging modality including echocardiography, CT, MRI, or angiography) who also have positive genetic testing results related to aortopathy.
- Aortic Valve Disease- Closed to enrollment: Subjects with aortic valve disease (bicuspid, unicuspid, or tricuspid disease)
- Family Members- Open to external enrollment: Family members of eligible subjects
  •Only family members of subjects with syndromic diagnoses are eligible for external enrollment at this time
- Controls- Closed to external enrollment: Control subjects having tissue removed during a surgical procedure (e.g. coronary artery bypass graft surgery (CABG), cardiac transplant, etc.)

SUMMARY:
The main purpose of this study is to define the complex genetic and pathogenic basis of thoracic aortic aneurysm (TAA) and other forms of aortopathy and/or aortic valve disease by identifying novel disease-causing genes and by identifying important genetic modifiers for aortic and aortic valve disease severity.

DETAILED DESCRIPTION:
Thoracic aortic aneurysm (TAA) is a type of aortopathy describing dilation of the proximal aortic dimensions including the aortic root, which is a risk factor for aortic dissection and sudden cardiac death. TAA and other forms of aortopathy (e.g. aortic tortuosity or aortic hypoplasia/stenosis) develop in the presence or absence of additional cardiovascular malformations including bicuspid aortic valve. TAA is associated with connective tissue disorders (e.g. Marfan syndrome), and familial clustering has been identified in a significant proportion of nonsyndromic cases, establishing high heritability. Pedigree analysis of TAA kindreds clearly identifies complex inheritance; however, progress towards understanding the genetic basis of TAA and other forms of aortopathy and, ultimately, the susceptibility to aortic dissection remains incomplete. There is a clinical need to develop novel methods for predicting disease risk based on genotype and phenotype, to further elucidate the genetic and pathogenic mechanisms of aortopathy, and to improve medical and surgical therapies. The overarching hypothesis of this study is that individual genetic variation modulates susceptibility to disease severity and progression. The goals of this study are 1) to ascertain a cohort of subjects who have aortopathy and/or aortic valve disease including TAA or who have genetic risk for the development of aortopathy and/or aortic valve disease, 2) to collect paired blood and tissue samples from well-characterized subjects, family members of subjects, and controls to perform genome-wide DNA sequence, histopathologic, transcriptional, and proteomic analyses, and 3) to establish a tissue biorepository with detailed phenotype information to facilitate a broad spectrum of current and future studies.

ELIGIBILITY:
Inclusion Criteria:

* Open to external enrollment:

  * Subjects with a genetic diagnosis of Marfan Syndrome (MDS), Loeys-Dietz Syndrome (LDS), or Vascular Ehlers-Danlos Syndrome (EDS); (Positive genetic testing or a previous cardiac study required to be eligible)
  * Family members of eligible subjects (Only family members of subjects with syndromic diagnoses are eligible for external enrollment at this time)
* Closed to external enrollment:

  * Subjects with aortic disease including TAA* or dissection, aortic tortuosity, or aortic hypoplasia/stenosis (based on any cardiac imaging modality including echocardiography, CT, MRI, or angiography)
  * Subjects with aortic valve disease (bicuspid, unicuspid, or tricuspid disease)
  * Control subjects having tissue removed during a surgical procedure (e.g. coronary artery bypass graft surgery (CABG), cardiac transplant, etc.)

Exclusion Criteria:

• Inability or unwillingness to provide consent (assent when indicated)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families affected by aortopathy, aortic valve disease, or syndromic or genetic diagnosis that poses risk for the development of aortic disease who have not yet developed disease.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-12-10; Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Biorepository Establishment | 20 years
  Establish a biorepository with detailed phenotype information to facilitate a broad spectrum of current and future studies
Genetic Analysis | 20 years
  The mechanisms of TAA pathogenesis will be determined by studying explanted aortic tissue and cells derived from patients with TAA for gene expression, protein expression, and other functional assays.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Landis, MD, Principal Investigator — IU School of Medicine
Locations (2):
- United States (2):
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - IU School of Medicine, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No